CLINICAL TRIAL: NCT03185832
Title: Heart Failure Indication and Sudden Cardiac Death Prevention Trial Japan
Brief Title: Heart Failure and Sudden Cardiac Death Japan Registry
Acronym: HINODE
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Other Study IDs: C2076
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Results first posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Heart Failure; Arrhythmias, Cardiac; Sudden Cardiac Death
Keywords: Hear failure; Sudden Cardiac Death; Arrhythmia; Implanted device; ICD; CRT
MeSH Terms: conditions — Heart Failure; Arrhythmias, Cardiac; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (4):
- CRT-D Cohort: Number of participants with first appropriately treated ventricular arrhythmia
  Interventions: Device: CRT-D
- ICD Cohort: Number of participants with first appropriately treated ventricular arrhythmia
  Interventions: Device: ICD
- Pacing (PM / CRT-P) Cohort: All cause mortality
  Interventions: Device: PM / CRT-P
- Non-device Cohort: All-cause mortality in the subject cohort with 2 to 5 predefined SCD driving risk factors
  Interventions: Other: Non-device

INTERVENTIONS:
Device: CRT-D — This subject cohort is made by all patients enrolled and implanted with defibrillator with CRT capabilities
  Groups: CRT-D Cohort
Device: ICD — This subject cohort is made by all patients enrolled and implanted with defibrillator capabilities
  Groups: ICD Cohort
Device: PM / CRT-P — This subject cohort is made by all patients enrolled and implanted with pacemakers with or without CRT capabilities
  Groups: Pacing (PM / CRT-P) Cohort
Other: Non-device — Patient enrolled but not implanted with a Defibrillator or Pacemaker
  Groups: Non-device Cohort

SUMMARY:
The purpose of this observational registry is to collect clinical events and outcome data in 4 different study populations (cohorts), with a majority of Japanese subjects, that are at risk of sudden cardiac death (SCD) and heart failure (HF) events. These event rates will be compared with available published data mainly from Europe and the United States.

Selected Subject Cohorts:

1. Selected subject cohort with criteria for SCD (without spontaneous prior ventricular sustained arrhythmia) and de novo Implantable Cardioverter-Defibrillator (ICD) device treatment.
2. Selected subject cohort with criteria for SCD and widely accepted standard cardiac resynchronization therapy (CRT) indication who received a de novo CRT-Defibrillator (CRT-D) device treatment.
3. Selected subject cohort who are clinically expected to require >40% right ventricular pacing with a left ventricular ejection fraction (LVEF) ≤50%, any determined New York Heart Association (NYHA) Class, and receiving pacemaker (PM) or CRT-Pacemaker (CRT-P) therapy despite previous device history (de novo, box changes, system revisions or upgrades).
4. Selected subject cohort with criteria for SCD fulfilling European Society of Cardiology (ESC) ICD or CRT-D therapy guidelines (2016) with an LVEF ≤35%, having 2 to 5 predefined SCD risk factors but do not have or had have a cardiac implanted defibrillator, CRT-D, PM, or CRT-P.

The primary endpoint will report on the Composite rate of first appropriately treated ventricular arrhythmia (by anti-tachycardia pacing [ATP] or shock) or life-threatening symptoms associated to ventricular arrhythmia (defined as hemodynamic instability which requires treatment), whichever comes first under MADIT RIT Arm B or C programming conditions in a study population with a majority of Japanese subjects. This primary end point is assessed in the ICD/CRT-D implanted patient cohort.

The all-cause mortality in subjects with a maximum of 3 risk factors (analyzed for MADIT II data) will be assessed in the Pacing (PM/CRT-P) patient cohort.

The all-cause mortality will be assessed in the non-implanted subject cohort.

ELIGIBILITY:
General Inclusion Criteria:

1. Subject is aged 20 or above
2. Subject is willing and capable of providing informed consent
3. Subject is willing and capable of participating in all visits associated with this study at an approved clinical study site and at the intervals defined by this Clinical Investigation Plan (CIP)
4. Measured Ejection fraction value obtained by echocardiography or equivalent method as Standard of Care (SOC):

   * Device cohorts: within the last 3 months prior to enrolment
   * Non-device cohort: latest available within the last 12 months prior to enrollment in case there was no documented HF decompensation, myocardial infarction (MI) or revascularization, otherwise within the last 3 months prior to enrollment

And 12 lead electrocardiogram (ECG) recording available as SOC:

* Device cohorts: pre-implant ECG maximum 45 days before implant; post-implant ECG
* Non-device cohort: latest available maximum 12 months prior to enrollment and subject agrees in the data being used for this study

General Exclusion Criteria:

1. Subject is enrolled in any other concurrent study without prior written approval from Boston Scientific (BSC), with the exception of local mandatory governmental registries and observational studies/registries that are not in conflict and do not affect the following:

   * Schedule of procedures for the HINODE Study (i.e. should not cause additional or missed visits)
   * HINODE Study outcome
   * Conduct of the HINODE Study per Good Clinical Practice /International Standard Organization 14155:2011/local regulations as applicable
2. Device implant revision is scheduled due to unstable result of an implant <45 days prior enrolment
3. Subjects with more than 5 of the following risk factors: LVEF <35%, NYHA Class III or IV, left bundle branch block (LBBB) with QRS > 130 ms or QRS ≥150 ms, renal dysfunction (chronically BUN >26 mg/dL / ≥9.28 mmol/L), diabetes type I and II, chronic atrial fibrillation (permanent or persistent according to ESC Guideline 2016), prior MI, age >70 years, smoking today or during last 5 years
4. Subjects with chronic renal disease with chronic BUN ≥50mg/dL or creatinine ≥2.5 mg/dL
5. Subjects with coronary artery bypass graft (CABG) surgery or percutaneous coronary intervention (PCI) within the past three calendar months prior to enrollment
6. Subjects with enzyme-positive myocardial infarction within the past three calendar months prior to enrollment
7. Subjects who are expected to survive for <1 year with good functional status
8. Subject's physician does not allow participation
9. Subject is not willing and capable of participating in all testing or visits associated with this clinical study at an approved clinical study center and at the intervals defined by this CIP
10. Unwilling to sign the consent for participation
11. Women of childbearing potential who are or might be pregnant at the time of study enrolment
12. ICD and CRT-D cohorts: implanted with a non-BSC device system. PM/CRT-P cohorts: implanted with a non-BSC pulse generator device.

Additional eligibility criteria apply to each cohort

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects enrolled in this observational registry are from the general population seen by enrolling physicians at primary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 354 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kazutaka Aonuma, Professor, Principal Investigator — University of Tsukuba Hospital
Locations (34):
- Japan (34):
  - Ichinomiya Municipal Hospital, Ichinomiya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Japanese Red Cross Nagoya Daini Hospital, Nagoya, Aichi-ken
  - Toho University Sakura Medical Center, Sakura, Chiba
  - Juntendo University Urayasu Hospital, Urayasu, Chiba
  - Fukuoka Tokushukai Hospital, Kasuga, Fukuoka
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Sapporo Higashi Tokushukai Hospital, Sapporo, Hokkaido
  - Kansai Rosai Hospital, Amagasaki, Hyōgo
  - Hyogo Brain and Heart Center, Himeji, Hyōgo
  - Hitachi General Hospital, Hitachi, Ibaraki
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - St. Marianna University School of Medicine Hospital, Kawasaki, Kanagawa
  - Yokohama Rosai Hospital, Yokohama, Kanagawa
  - Yokohama Minami Kyousai Hospital, Yokohama, Kanagawa
  - St. Marianna University School of Medicine, Yokohama City Seibu Hospital, Yokohama, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - National Cerebral and Cardiovascular Center Hospital, Suita, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Tokyo Medical and Dental University Medical Hospital, Bunkyo, Tokyo
  - Nippon Medical School Hospital, Bunkyō, Tokyo
  - St. Luke's International Hospital, Chūō, Tokyo
  - Toho University Ohashi Medicine Center, Meguro City, Tokyo
  - Toho University Omori Medical Center, Ōta-ku, Tokyo
  - Tokyo Metropolitan Hiroo Hospital, Shibuya City, Tokyo
  - Yamaguchi University Hospital, Ube, Yamaguchi
  - Kokura Memorial Hospital, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Okayama University Hospital, Okayama
  - Sakurabashi Watanabe Hospital, Osaka
  - Osaka General Medical Center, Osaka
  - Jichi Medical University Saitama Medical Center, Saitama
  - Japanese Red Cross Saitama Hospital, Saitama

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled on 21 July 2017 and the last subject follow-up occurred on 14 September 2020. Study completion date, defined as the date the final participant was examined or received an intervention for purposes of final collection of data for the primary and secondary outcome measures and adverse events, is 1 December 2020. A total of 354 subjects across 34 centers in Japan were enrolled and assigned to a study cohort.
Pre-assignment Details: Out of 357 enrolled patients, 3 did not meet eligibility criteria and were considered consent ineligible.
Groups:
- CRT-D Cohort: This subject cohort is made by all patients enrolled and implanted with cardiac resynchronization therapy defibrillator (CRT-D)
- ICD Cohort: This subject cohort is made by all patients enrolled and implanted with implantable cardioverter-defibrillator (ICD)
- Pacing Cohort: This subject cohort is made by all patients enrolled and implanted with pacemakers (PM) with or without cardiac resynchronization therapy (CRT) capabilities
- Non-device Cohort: Patient enrolled but not implanted with a Defibrillator or Pacemaker
Period: Overall Study
Arm/Group | CRT-D Cohort | ICD Cohort | Pacing Cohort | Non-device Cohort
Started | 69 | 102 | 68 | 115
Completed | 60 | 87 | 58 | 104
Not Completed | 9 | 15 | 10 | 11
Not completed — Death | 9 | 14 | 9 | 7
Not completed — Withdrawn - vital status available | 0 | 1 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- CRT-D Cohort: This subject cohort is made by all patients enrolled and implanted with defibrillator with CRT capabilities
- ICD Cohort: This subject cohort is made by all patients enrolled and implanted with defibrillator capabilities
- Pacing Cohort: This subject cohort is made by all patients enrolled and implanted with pacemakers with or without CRT capabilities
- Total: Total of all reporting groups
Arm/Group | CRT-D Cohort | ICD Cohort | Pacing Cohort | Non-device Cohort | Total
Number analyzed (Participants) | 69 | 102 | 68 | 115 | 354
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (13.4) | 68.2 (10.4) | 75.0 (10.9) | 68.8 (11.8) | 69.4 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 15 | 24 | 25 | 86
  Male | 47 | 87 | 44 | 90 | 268
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Japan | 69 | 102 | 68 | 115 | 354

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Ventricular Arrhythmia Associated Symptoms - ICD/CRT-D Cohorts
Description: Number of Participants with first appropriately treated ventricular arrhythmia (by anti tachycardia pacing [ATP] or shock) or life-threatening symptoms associated to ventricular arrhythmia (defined as hemodynamic instability which requires treatment), whichever comes first under MADIT Arm B or C programming conditions in a study population with a majority of Japanese subjects.
Time Frame: 12 months follow up
Population: ICD Cohort: subjects with criteria for sudden cardiac death (SCD) (without spontaneous prior ventricular sustained arrhythmia) and de novo implanted Defibrillator device treatment (ICD).
  CRT-D Cohort: subjects with criteria for SCD and widely accepted standard CRT indication who received a de novo implanted CRT D device treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | CRT-D Cohort | ICD Cohort
Number analyzed (Participants) | 69 | 102
Participants | 3 | 8

2. Primary Outcome: Number of Participant Deaths - Pacing Cohort
Description: All-cause mortality in subjects with a maximum of 3 risk factors (analyzed for MADIT II data).
Time Frame: 12 months follow up
Population: Subjects who were clinically expected to require >40% right ventricular pacing with a left ventricular ejection fraction (LVEF) ≤50%, any determined New York Heart Association (NYHA) Class, and receiving PM or CRT-Pacemaker (CRT-P) therapy despite previous device history (de novo, box changes, system revisions or upgrades).
Measure: Count of Participants; unit: Participants
Arm/Group | Pacing Cohort
Number analyzed (Participants) | 39
Participants | 3

3. Primary Outcome: Number of Participant Deaths - Non-Device Cohort
Description: All-cause mortality in the subject cohort with 2 to 5 predefined SCD driving risk factors.
Time Frame: 12 months follow up
Population: Subjects with criteria for SCD fulfilling European Society of Cardiology (ESC) ICD or CRT-D therapy guidelines (2016) with an LVEF ≤35%, having 2 to 5 predefined risk factors but do not have or have had a cardiac implanted device ICD, CRT-D, PM, or CRT-P.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-device Cohort
Number analyzed (Participants) | 115
Participants | 5

4. Secondary Outcome: Number of Participant Deaths - ICD/CRT-D Cohorts
Description: All-cause mortality for the ICD and the CRT-D cohorts.
Time Frame: 12 months follow up
Population: ICD Cohort: subjects with criteria for SCD (without spontaneous prior ventricular sustained arrhythmia) and de novo implanted Defibrillator device treatment (ICD).
  CRT-D Cohort: subject with criteria for SCD and widely accepted standard CRT indication who received a de novo implanted CRT D device treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | CRT-D Cohort | ICD Cohort
Number analyzed (Participants) | 69 | 102
Participants | 5 | 3

5. Secondary Outcome: Number of Participants With Composite HF Event - ICD/CRT-D/Pacing Cohorts
Description: Number of Participants with HF events, which require intravenous (IV) treatment and/or heart failure (HF) related hospitalization, or which led to HF death
Time Frame: 12 months follow up
Population: ICD Cohort: subjects with criteria for SCD (without spontaneous prior ventricular sustained arrhythmia) and de novo ICD implant.
  CRT-D Cohort: subject with criteria for SCD and widely accepted standard CRT indication who received a de novo CRT-D implant.
  PM/CRT-P Cohort: subjects who were clinically expected to require >40% right ventricular pacing with an LVEF ≤50%, any determined New York Heart Association (NYHA) Class, and receiving PM or CRT-P therapy despite previous device history.
Measure: Count of Participants; unit: Participants
Arm/Group | CRT-D Cohort | ICD Cohort | Pacing Cohort
Number analyzed (Participants) | 69 | 102 | 68
Participants | 16 | 27 | 9

6. Secondary Outcome: Number of Participants With Complication - ICD/CRT-D/Pacing Cohorts
Description: Complication refers to qualified serious adverse device effects (SADEs) post success implantation, such as re-implant procedure, required invasive procedure related to the device system, pacing exit block, all-cause infection, and death due to therapy failure.
Time Frame: 12 months follow up
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | CRT-D Cohort | ICD Cohort | Pacing Cohort
Number analyzed (Participants) | 69 | 102 | 68
Participants | 3 | 4 | 2

ADVERSE EVENTS:
Time Frame: Adverse events are collected through study completion, an average of 20 months
Description: All adverse events are collected as per ISO 14155 and medical device guidance (MEDDEV) 2.7/4.
  As per protocol, adverse events were collected irrespective of cohort allocation and therefore are not reported separately
Groups:
- Actively Enrolled Patients: Patients actively enrolled in the study, defined as subjects who met all eligibility criteria and who signed informed consent
Arm/Group | Actively Enrolled Patients
All-Cause Mortality (participants affected / at risk) | 39/354
Serious Adverse Events (participants affected / at risk) | 172/354
Other Adverse Events (participants affected / at risk) | 99/354
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Actively Enrolled Patients (N=354)
Infection (> 30 days post implant) (Product Issues) | 2/239 (2)
Hematoma- Pocket (>30 days post implant) (Surgical and medical procedures) | 1/239 (1)
Elevated Threshold - RV Lead (Product Issues) | 2/171 (2)
Elevated Threshold - LV Lead (Product Issues) | 1/115 (1)
Post-surgical pocket hemorrhage/bleeding/drainage (Surgical and medical procedures) | 2/239 (2)
Post -Surgical infection (<= 30 days post implant) (Surgical and medical procedures) | 1/239 (1)
Hematoma - pocket (<= 30 days post-implant) (Surgical and medical procedures) | 2/239 (2)
Syncope - Heart Failure (Cardiac disorders) | 1 (1)
Dizziness - Heart Failure (Cardiac disorders) | 1 (1)
Chest Pain - Heart Failure (Cardiac disorders) | 1 (1)
Dyspnea - Heart Failure (Cardiac disorders) | 38 (46)
Peripheral edema - Heart Failure (Cardiac disorders) | 2 (8)
Fatigue - Heart Failure (Cardiac disorders) | 5 (5)
Renal Failure/Insufficiency - Heart Failure (Renal and urinary disorders) | 3 (3)
Dehydration - Heart Failure (Cardiac disorders) | 1 (1)
Weight Gain - Heart Failure (Cardiac disorders) | 4 (4)
Pleural Effusion - Heart Failure (Cardiac disorders) | 1 (1)
Cardiac Medication Complication - Heart Failure (Cardiac disorders) | 1 (1)
Heart Failure Symptoms - Unspecified (Cardiac disorders) | 21 (23)
Multiple Heart Failure Symptoms (Cardiac disorders) | 28 (35)
Other - Heart failure patient condition (Cardiac disorders) | 4 (4)
Sinus Bradycardia (Cardiac disorders) | 1 (1)
Ventricular Fibrillation (VF) (Cardiac disorders) | 6 (6)
Ventricular Tachycardia (VT)/Monomorphic VT (Cardiac disorders) | 13 (22)
Nonsustained ventricular tachycardia (NSVT) (Cardiac disorders) | 1 (1)
Atrial Fibrillation (AF) (Cardiac disorders) | 13 (14)
Atrial Flutter (Cardiac disorders) | 1 (1)
Atrial Tachycardia/Other SVT (e.g. AVRT, AVNRT, EAT) (Cardiac disorders) | 3 (3)
Premature Ventricular Contractions (PVC) (Cardiac disorders) | 2 (2)
Cardiac Arrest (Cardiac disorders) | 2 (2)
Myocardial Infarction (Cardiac disorders) | 2 (2)
Coronary Artery Disease (Cardiac disorders) | 7 (8)
Peripheral Vascular Disease (General disorders) | 4 (4)
Mitral Regurgitation (Cardiac disorders) | 3 (3)
Tricuspid Regurgitation (Cardiac disorders) | 1 (1)
Dizziness (Cardiac disorders) | 1 (1)
Chest Pain - Ischemic (Cardiac disorders) | 6 (6)
Chest Pain - Other (Cardiac disorders) | 2 (2)
Other - Patient condition (General disorders) | 5 (5)
Transient Ischemic Attack (TIA) (Nervous system disorders) | 1 (1)
Cerebrovascular Accident (CVA) (Nervous system disorders) | 2 (2)
Cerebrovascular accident (CVA) - ischemic (Nervous system disorders) | 1 (1)
Pneumothorax - unrelated procedure/device (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other - Unrelated to procedure/device (General disorders) | 1 (1)
Adverse Reaction - Medication (General disorders) | 4 (4)
Other - Patient condition (General disorders) | 2 (2)
Death (General disorders) | 7 (7)
System Infection (Product Issues) | 2 (2)
Fever and/or Virus (General disorders) | 1 (1)
Physical Trauma (General disorders) | 9 (9)
Localized Infection (General disorders) | 1 (1)
Hematological (Blood and lymphatic system disorders) | 1 (1)
Neurological (Nervous system disorders) | 4 (4)
Gastrointestinal (Gastrointestinal disorders) | 12 (15)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 16 (16)
Other - Whole body (General disorders) | 2 (3)
Genitourinary (Reproductive system and breast disorders) | 3 (3)
Renal (Renal and urinary disorders) | 4 (4)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 5 (5)
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 4 (4)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (15)
Incisional/Superficial Infection (<= 30d post implant without explant) (Product Issues) | 1/16 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Actively Enrolled Patients (N=354)
Extracardiac Stimulation - LV PG System (Product Issues) | 1/239 (1)
Inappropriate tachy therapy - SVT - Defibrillation Lead (Product Issues) | 3/171 (3)
Extracardiac Stimulation - LV Lead (Product Issues) | 3/115 (4)
Hematoma - pocket (<= 30 days post-implant) (Product Issues) | 1/239 (1)
Dizziness - Heart Failure (Cardiac disorders) | 1 (1)
Chest Pain - Heart Failure (Cardiac disorders) | 1 (1)
Dyspnea - Heart Failure (Cardiac disorders) | 12 (14)
Renal Failure/Insufficiency - Heart Failure (Renal and urinary disorders) | 1 (1)
Dehydration - Heart Failure (Cardiac disorders) | 1 (1)
Heart Failure Symptoms - Unspecified (Cardiac disorders) | 5 (5)
Multiple Heart Failure Symptoms (Cardiac disorders) | 6 (6)
Other - Heart failure patient condition (Cardiac disorders) | 2 (2)
Ventricular Fibrillation (VF) (Cardiac disorders) | 3 (3)
Ventricular Tachycardia (VT)/Monomorphic VT (Cardiac disorders) | 11 (46)
Nonsustained ventricular tachycardia (NSVT) (Cardiac disorders) | 2 (2)
Atrial Fibrillation (AF) (Cardiac disorders) | 14 (15)
Atrial Flutter (Cardiac disorders) | 1 (1)
Atrial Tachycardia/Other SVT (e.g. AVRT, AVNRT, EAT) (Cardiac disorders) | 3 (3)
Hypotension/Orthostatic Hypotension (Cardiac disorders) | 1 (1)
Hypertension/Hypertensive Crisis (Cardiac disorders) | 1 (1)
Mitral Regurgitation (Cardiac disorders) | 1 (1)
Syncope (Cardiac disorders) | 1 (1)
Dizziness (Cardiac disorders) | 3 (4)
Dyspnea (Cardiac disorders) | 2 (2)
Other - Patient condition (General disorders) | 1 (1)
Transient Ischemic Attack (TIA) (Nervous system disorders) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1)
Hemorrhage - unrelated procedure/device (General disorders) | 1 (1)
Pleural Effusion - unrelated procedure/device (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Adverse Reaction - Medication (General disorders) | 2 (2)
System Infection (Product Issues) | 1 (1)
Fever and/or Virus (General disorders) | 5 (5)
Physical Trauma (General disorders) | 9 (10)
Hematological (Blood and lymphatic system disorders) | 2 (2)
Neurological (Nervous system disorders) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 5 (5)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Genitourinary (Reproductive system and breast disorders) | 1 (1)
Renal (Renal and urinary disorders) | 24 (30)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 2 (2)
Integumentary (Skin and subcutaneous tissue disorders) | 1 (3)
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 4 (4)
Endocrine (Endocrine disorders) | 2 (2)
Inappropriate Tachy Therapy - Other - PG (Product Issues) | 1/16 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-29): https://cdn.clinicaltrials.gov/large-docs/32/NCT03185832/Prot_SAP_000.pdf